CLINICAL TRIAL: NCT03912935
Title: Comparison of Bed up Head Elevated Position With Sniffing Position in Rapid Sequence Induction: a Randomised, Controlled, Non-inferiority Trial
Brief Title: Comparison of Bed up Head Elevated Position With Sniffing Position in Rapid Sequence Induction.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Shahmini a/p Ganesh, Principal Investigator, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MREC ID NO: 2018222-6042
Record Dates: First submitted 2019-03-09; First posted 2019-04-11 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Endotracheal Intubation in Bed up Head Elevation Position in Rapid Sequence Induction
Keywords: Rapid sequence induction; Bed up head elevation; sniffing position; cricoid pressure; time taken for intubation in seconds; percentage of glottic opening

STUDY DESIGN:
Intervention Model Description: * All patients undergoing elective surgery under general anaesthesia from age 18 years old to 75 years old selected.
  * Written informed consent will be obtained prior to enrolment.
  * Randomisation into 2 groups (BUHE and sniffing position) will be done via computer generated sequences. Subsequently, will be placed into sealed envelopes.
  * The next available envelope will be selected and open for that particular patient at the time of enrolment.
Who Masked: Participant
Masking Description: Only participant is masked from knowing the assigned group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sniffing position (No Intervention): Subject will be maintained in standard intubation position which is supine position with head elevation with head rest (foam donut).
- Bed up head elevation position (Experimental): Subject will be maintained at bed up 20-30 degree aiming alignment between the external auditory meatus with sternal notch
  Interventions: Other: comparison between two different intubating position

INTERVENTIONS:
Other: comparison between two different intubating position — Comparing to different position (sniffing and BUHE) in endotracheal intubation for rapid sequence induction in simulated emergency cases
  Arms: Bed up head elevation position

SUMMARY:
This study is aimed to conduct a randomised controlled trial comparing endotracheal intubation (ETI) in bed up head elevation BUHE position versus sniffing position in simulated rapid sequence induction (RSI).

Objective is to determine if the time taken for intubation in the bed up head elevated position is non-inferior to time taken for intubation in the sniffing position.

The hypotheses:

1. In patients undergoing rapid sequence induction in simulated emergency surgery under general anaesthesia, direct laryngoscopy (DL) and ETI in the BUHE position is non inferior to time required for DL and successful ETI in the sniffing position.
2. In patients undergoing rapid sequence induction in simulated emergency surgery under general anaesthesia, direct laryngoscopy (DL) and ETI in the BUHE position improve POGO score.
3. In patients undergoing rapid sequence induction in simulated emergency surgery under general anaesthesia, direct laryngoscopy (DL) and ETI in the BUHE position reduces airway related complications.

Terminology:

Direct laryngoscopy (DL) and Endotracheal intubation (ETI): Is a method of inserting a breathing tube into the trachea (windpipe) once patient undergo general anaesthesia.

Bed up head elevation (BUHE): Bed up at 20-30 degree aiming alignment between the external auditory meatus with sternal notch.

Sniffing position: Maintaining supine position with head elevation with head rest.

Rapid sequence induction (RSI): An established method of inducing anaesthesia in patients who are at risk of aspiration of gastric contents into the lungs. It involves loss of consciousness during cricoid pressure followed by intubation without face mask ventilation. The aim is to intubate the trachea as quickly and as safely as possible.

POGO score: Percentage of glottic opening

Cricoid Pressure (CP): Maneuvre to prevent regurgitation of gastric contents during induction of anaesthesia by temporary occlusion of the upper end of the esophagus by backward pressure of cricoid cartilage against bodies of cervical vertebrae.

DETAILED DESCRIPTION:
All patients from age 18 years old to 75 years old undergoing elective surgery under general anaesthesia in operating theater of University Malaya Medical Centre over a period of 15 months, from April 2018 to June 2019 will be included and recruited based on inclusion and exclusion criteria.

Those patient that fulfilled the criteria and consented for the study will be randomized to 2 group.

i) BUHE group: Bed up at 20-30 degree aiming alignment between the external auditory meatus with sternal notch.

ii) Sniffing group: Maintaining supine position with head elevation with head rest (foam donut).

Induction of anaesthesia starts with:

* preoxygenation with 100% oxygen for 3-5 min performed until end tidal oxygen of 85% achieved.
* A pre-calculated dose of induction agent is administered, followed immediately by a neuromuscular blocking agent.

(IV Fentanyl 2mcg/kg,IV Propofol 2-3mg/kg,IV Rocuronium 1mg/kg).

* Cricoid pressure at 10 Newton is applied increasing to 30 Newton once consciousness is lost.
* After adequate neuromuscular blockade,both group patients will be intubated by one investigator via direct laryngoscopy using Macintosh blade size 3 or 4.
* Time taken from insertion of Macintosh blade into oral cavity till confirmation of endotracheal tube placement via detection of CO2 on the end tidal CO2 monitor will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing elective surgery under general anaesthesia from age 18 years old to 75 years old.

Exclusion Criteria:

* Patients with airway obstruction
* Patients with contraindication to neck extension
* BMI> 35kg/m2
* Patient with history of difficult airway from previous intubation history
* Only single intubation will be included if patients had multiple surgery during their hospital stay
* Patients with ischaemic heart disease, cerebrovascular diseases and respiratory disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2018-08-24 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Time in seconds measured from when the laryngoscopy blade passes through the incisors to the first measured end tidal CO2 wave | Intraoperatively , during induction of anaesthesia
  Measured from when the laryngoscopy blade passes through the incisors to the first measured end tidal CO2 wave

SECONDARY OUTCOMES:
Number of laryngoscopy and intubation attempt | Intraoperatively , during induction of anaesthesia
  Number of attempts taken by investigator to obtain successful endotracheal intubation in both arms
Laryngeal exposure measured via POGO score | Intraoperatively , during induction of anaesthesia
  Percentage of glottic opening during laryngoscopy
Occurrence of difficult intubation | Intraoperatively , during induction of anaesthesia
  Defined as ≥3 attempts at intubation
Occurrence of hypoxia | Intraoperatively , during induction of anaesthesia
  Hypoxia defined as pulse oximetry reading less than 95 percents
The use of any other airway adjunct or external laryngeal manipulation to assist in intubation | Intraoperatively , during induction of anaesthesia
  Change of blade size, bougie, magill forcep, video assisted laryngoscope,external laryngeal manipulation (Use of any airway adjunct is grouped as one)
Occurrence of esophageal intubation | Intraoperatively , during induction of anaesthesia
  Unsuccessful intubation into esophagus
Occurrence of airway trauma | Intraoperatively , during induction of anaesthesia
  broken tooth, bleeding or injury from oral cavity, tongue or lips, etc

CONTACTS AND LOCATIONS:
Overall Officials: Shahmini Ganesh, MD, Principal Investigator — UMMC
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data that already summarized and analysed in the form of schematic diagram will be available to other researchers

REFERENCES:
- [Background] Brodsky JB. Positioning the morbidly obese patient for anesthesia. Obes Surg. 2002 Dec;12(6):751-8. doi: 10.1381/096089202320995510. PMID 12568178
- [Background] SELLICK BA. Cricoid pressure to control regurgitation of stomach contents during induction of anaesthesia. Lancet. 1961 Aug 19;2(7199):404-6. doi: 10.1016/s0140-6736(61)92485-0. No abstract available. PMID 13749923
- [Background] Vanner RG, Pryle BJ. Nasogastric tubes and cricoid pressure. Anaesthesia. 1993 Dec;48(12):1112-3. doi: 10.1111/j.1365-2044.1993.tb07560.x. No abstract available. PMID 8068068
- [Background] Smith KJ, Ladak S, Choi PT, Dobranowski J. The cricoid cartilage and the esophagus are not aligned in close to half of adult patients. Can J Anaesth. 2002 May;49(5):503-7. doi: 10.1007/BF03017931. PMID 11983669
- [Background] Rice MJ, Mancuso AA, Gibbs C, Morey TE, Gravenstein N, Deitte LA. Cricoid pressure results in compression of the postcricoid hypopharynx: the esophageal position is irrelevant. Anesth Analg. 2009 Nov;109(5):1546-52. doi: 10.1213/ane.0b013e3181b05404. PMID 19843793
- [Background] Robinson JS, Thompson JM. Fatal aspiration (Mendelson's) syndrome despite antacids and cricoid pressure. Lancet. 1979 Aug 4;2(8136):228-30. doi: 10.1016/s0140-6736(79)90240-x. PMID 89335
- [Background] Williamson R. Cricoid pressure. Can J Anaesth. 1989 Sep;36(5):601. doi: 10.1007/BF03005396. No abstract available. PMID 2791184
- [Background] Kluger MT, Short TG. Aspiration during anaesthesia: a review of 133 cases from the Australian Anaesthetic Incident Monitoring Study (AIMS). Anaesthesia. 1999 Jan;54(1):19-26. doi: 10.1046/j.1365-2044.1999.00642.x. PMID 10209365
- [Background] Schwartz DE, Matthay MA, Cohen NH. Death and other complications of emergency airway management in critically ill adults. A prospective investigation of 297 tracheal intubations. Anesthesiology. 1995 Feb;82(2):367-76. doi: 10.1097/00000542-199502000-00007. PMID 7856895
- [Background] Thibodeau LG, Verdile VP, Bartfield JM. Incidence of aspiration after urgent intubation. Am J Emerg Med. 1997 Oct;15(6):562-5. doi: 10.1016/s0735-6757(97)90157-1. PMID 9337361
- [Background] Tomkinson J, Turnbull A, Robson G, Cloake E, Adelstein AM, Weatherall J. Report on confidential enquiries into maternal deaths in England and Wales 1973-1975. Rep Health Soc Subj (Lond). 1979;14:1-166. No abstract available. PMID 493710
- [Background] Guirro UB, Martins CR, Munechika M. Assessment of anesthesiologists' rapid sequence induction technique in an university hospital. Rev Bras Anestesiol. 2012 May-Jun;62(3):335-45. doi: 10.1016/S0034-7094(12)70134-4. PMID 22656679
- [Background] Schmidt A, Akeson J. Practice and knowledge of cricoid pressure in southern Sweden. Acta Anaesthesiol Scand. 2001 Nov;45(10):1210-4. doi: 10.1034/j.1399-6576.2001.451006.x. PMID 11736671
- [Background] Brimacombe J, White A, Berry A. Effect of cricoid pressure on ease of insertion of the laryngeal mask airway. Br J Anaesth. 1993 Dec;71(6):800-2. doi: 10.1093/bja/71.6.800. PMID 8280541
- [Background] Vanner RG, Clarke P, Moore WJ, Raftery S. The effect of cricoid pressure and neck support on the view at laryngoscopy. Anaesthesia. 1997 Sep;52(9):896-900. doi: 10.1111/j.1365-2044.1997.181-az0315.x. PMID 9349075
- [Background] Turgeon AF, Nicole PC, Trepanier CA, Marcoux S, Lessard MR. Cricoid pressure does not increase the rate of failed intubation by direct laryngoscopy in adults. Anesthesiology. 2005 Feb;102(2):315-9. doi: 10.1097/00000542-200502000-00012. PMID 15681945
- [Background] Adnet F, Racine SX, Borron SW, Clemessy JL, Fournier JL, Lapostolle F, Cupa M. A survey of tracheal intubation difficulty in the operating room: a prospective observational study. Acta Anaesthesiol Scand. 2001 Mar;45(3):327-32. doi: 10.1034/j.1399-6576.2001.045003327.x. PMID 11207469
- [Background] Magill IW. TECHNIQUE IN ENDOTRACHEAL ANAESTHESIA. Br Med J. 1930 Nov 15;2(3645):817-9. doi: 10.1136/bmj.2.3645.817. No abstract available. PMID 20775829
- [Background] Horton WA, Fahy L, Charters P. Defining a standard intubating position using "angle finder". Br J Anaesth. 1989 Jan;62(1):6-12. doi: 10.1093/bja/62.1.6. PMID 2917111
- [Background] Isono S. Common practice and concepts in anesthesia: time for reassessment: is the sniffing position a "gold standard" for laryngoscopy? Anesthesiology. 2001 Oct;95(4):825-7. doi: 10.1097/00000542-200110000-00007. No abstract available. PMID 11605919
- [Background] Akhtar M, Ali Z, Hassan N, Mehdi S, Wani GM, Mir AH. A Randomized Study Comparing the Sniffing Position with Simple Head Extension for Glottis Visualization and Difficulty in Intubation during Direct Laryngoscopy. Anesth Essays Res. 2017 Jul-Sep;11(3):762-766. doi: 10.4103/0259-1162.204206. PMID 28928584
- [Background] Brodsky JB, Lemmens HJ, Brock-Utne JG, Vierra M, Saidman LJ. Morbid obesity and tracheal intubation. Anesth Analg. 2002 Mar;94(3):732-6; table of contents. doi: 10.1097/00000539-200203000-00047. PMID 11867407
- [Background] Collins JS, Lemmens HJ, Brodsky JB, Brock-Utne JG, Levitan RM. Laryngoscopy and morbid obesity: a comparison of the "sniff" and "ramped" positions. Obes Surg. 2004 Oct;14(9):1171-5. doi: 10.1381/0960892042386869. PMID 15527629
- [Background] Lebowitz PW, Shay H, Straker T, Rubin D, Bodner S. Shoulder and head elevation improves laryngoscopic view for tracheal intubation in nonobese as well as obese individuals. J Clin Anesth. 2012 Mar;24(2):104-8. doi: 10.1016/j.jclinane.2011.06.015. Epub 2012 Feb 1. PMID 22301204
- [Background] Lee BJ, Kang JM, Kim DO. Laryngeal exposure during laryngoscopy is better in the 25 degrees back-up position than in the supine position. Br J Anaesth. 2007 Oct;99(4):581-6. doi: 10.1093/bja/aem095. Epub 2007 Jul 4. PMID 17611252
- [Background] Turner JS, Ellender TJ, Okonkwo ER, Stepsis TM, Stevens AC, Eddy CS, Sembroski EG, Perkins AJ, Cooper DD. Cross-over study of novice intubators performing endotracheal intubation in an upright versus supine position. Intern Emerg Med. 2017 Jun;12(4):513-518. doi: 10.1007/s11739-016-1481-z. Epub 2016 Jun 14. PMID 27300036
- [Background] Semler MW, Janz DR, Russell DW, Casey JD, Lentz RJ, Zouk AN, deBoisblanc BP, Santanilla JI, Khan YA, Joffe AM, Stigler WS, Rice TW; Check-UP Investigators( *); Pragmatic Critical Care Research Group. A Multicenter, Randomized Trial of Ramped Position vs Sniffing Position During Endotracheal Intubation of Critically Ill Adults. Chest. 2017 Oct;152(4):712-722. doi: 10.1016/j.chest.2017.03.061. Epub 2017 May 6. PMID 28487139
- [Background] Reddy RM, Adke M, Patil P, Kosheleva I, Ridley S; Anaesthetic Department at Glan Clwyd Hospital. Comparison of glottic views and intubation times in the supine and 25 degree back-up positions. BMC Anesthesiol. 2016 Nov 16;16(1):113. doi: 10.1186/s12871-016-0280-4. PMID 27852241
- [Background] El-Orbany MI, Getachew YB, Joseph NJ, Salem MR, Friedman M. Head elevation improves laryngeal exposure with direct laryngoscopy. J Clin Anesth. 2015 Mar;27(2):153-8. doi: 10.1016/j.jclinane.2014.09.012. Epub 2014 Nov 22. PMID 25468586
- [Background] Levitan RM, Mechem CC, Ochroch EA, Shofer FS, Hollander JE. Head-elevated laryngoscopy position: improving laryngeal exposure during laryngoscopy by increasing head elevation. Ann Emerg Med. 2003 Mar;41(3):322-30. doi: 10.1067/mem.2003.87. PMID 12605198
- [Background] Rao SL, Kunselman AR, Schuler HG, DesHarnais S. Laryngoscopy and tracheal intubation in the head-elevated position in obese patients: a randomized, controlled, equivalence trial. Anesth Analg. 2008 Dec;107(6):1912-8. doi: 10.1213/ane.0b013e31818556ed. PMID 19020138
- [Background] Turner JS, Ellender TJ, Okonkwo ER, Stepsis TM, Stevens AC, Sembroski EG, Eddy CS, Perkins AJ, Cooper DD. Feasibility of upright patient positioning and intubation success rates At two academic EDs. Am J Emerg Med. 2017 Jul;35(7):986-992. doi: 10.1016/j.ajem.2017.02.011. Epub 2017 Feb 5. PMID 28202295
- [Background] Hastings RH, Kelley SD. Neurologic deterioration associated with airway management in a cervical spine-injured patient. Anesthesiology. 1993 Mar;78(3):580-3. doi: 10.1097/00000542-199303000-00022. No abstract available. PMID 8457057
- [Background] Khandelwal N, Khorsand S, Mitchell SH, Joffe AM. Head-Elevated Patient Positioning Decreases Complications of Emergent Tracheal Intubation in the Ward and Intensive Care Unit. Anesth Analg. 2016 Apr;122(4):1101-7. doi: 10.1213/ANE.0000000000001184. PMID 26866753
- [Background] Dixon BJ, Dixon JB, Carden JR, Burn AJ, Schachter LM, Playfair JM, Laurie CP, O'Brien PE. Preoxygenation is more effective in the 25 degrees head-up position than in the supine position in severely obese patients: a randomized controlled study. Anesthesiology. 2005 Jun;102(6):1110-5; discussion 5A. doi: 10.1097/00000542-200506000-00009. PMID 15915022
- [Background] Boyce JR, Ness T, Castroman P, Gleysteen JJ. A preliminary study of the optimal anesthesia positioning for the morbidly obese patient. Obes Surg. 2003 Feb;13(1):4-9. doi: 10.1381/096089203321136511. PMID 12630606
- [Background] Sun DA, Warriner CB, Parsons DG, Klein R, Umedaly HS, Moult M. The GlideScope Video Laryngoscope: randomized clinical trial in 200 patients. Br J Anaesth. 2005 Mar;94(3):381-4. doi: 10.1093/bja/aei041. Epub 2004 Nov 26. PMID 15567809